CLINICAL TRIAL: NCT03722446
Title: A Head-to-head Comparison of Catheter Thread Between Two Epidural Kit Vendors.
Brief Title: Epidural Catheter Thread Between Two Different Vendors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Carlo Pancaro, Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 00143333
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arrow Catheter Kit. (Other): Arrow FlexTip Plus Epidural Catheterization Kit is a single orifice flex tip catheter used to place epidurals in pregnant women in labor who request an epidural for pain management in labor. This kit will be used in half of the randomized weeks.
  Interventions: Device: Arrow Catheter Kit.
- B.Braun Catheter Kit (Other): Perifix FX Springwound Epidural Catheter Kit is a multi-orifice flex tip catheter used to place epidurals in pregnant women in labor who request an epidural for pain management in labor. This kit will be used in half of the randomized weeks.
  Interventions: Device: B.Braun Catheter Kit

INTERVENTIONS:
Device: Arrow Catheter Kit. — The group will be randomized to receive this labor analgesia kit.
  Arms: Arrow Catheter Kit.
Device: B.Braun Catheter Kit — The group will be randomized to receive this labor analgesia kit.
  Arms: B.Braun Catheter Kit

SUMMARY:
The aim of the study is to assess if there is a difference in ability to thread the epidural catheter from two different epidural pain management kits vendors

DETAILED DESCRIPTION:
The aim of the study is to assess if there is a difference in ability to thread the epidural catheter from two different pain management kits. In order to improve patient care, if there is a difference in the time to thread epidurals with one kit over the other, we would like to use the kit with decreased time to thread in the future.

ELIGIBILITY:
Inclusion Criteria: women in labor

-

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pancaro, MD, Principal Investigator — University of Michigan
Locations (1):
- von Voitlander Women's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year

REFERENCES:
- [Derived] Pancaro C, Purtell J, LaBuda D, Saager L, Klumpner TT, Dubovoy T, Rajala B, Singh S, Cassidy R, Vahabzadeh C, Maxwell S, Manica V, Eckmann DM, Mhyre JM, Engoren MC. Difficulty in Advancing Flexible Epidural Catheters When Establishing Labor Analgesia: An Observational Open-Label Randomized Trial. Anesth Analg. 2021 Jul 1;133(1):151-159. doi: 10.1213/ANE.0000000000005526. PMID 33835077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in labor requesting epidural analgesia for an expected vaginal delivery.
Pre-assignment Details: Participants were excluded if there was a fetal loss involved.
Period: Overall Study
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Started | 135 | 122
Completed | 120 | 120
Not Completed | 15 | 2
Not completed — Protocol Violation | 15 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5) | 30 (6) | 30 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 120 | 240
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational Age [Mean (Standard Deviation); unit: weeks] | 38.9 (1.5) | 38.6 (2.6) | 38.8 (2.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (5.6) | 31.6 (6.7) | 31.6 (6.2)
Cervical Dilation [Mean (Standard Deviation); unit: cm] | 4 (2) | 4 (2) | 4 (2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Successful Thread at First Pass
Description: A thread is considered successful at first pass if there were no minor or major manipulations required.
Time Frame: within 60min of first attempt at placement
Measure: Count of Participants; unit: Participants
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
Participants | 81 | 117
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p < 0.0001, Chi-squared

2. Secondary Outcome: Time to Thread Epidural Catheter
Description: At the epidural placement, total amount of time required to establish successful epidural catheter thread
Time Frame: within 60min of first attempt at placement
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
seconds | 135 (186) | 51 (31)
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p = 0.01020, t-test, 1 sided

3. Secondary Outcome: Incidence of Unintended Dural Punctures
Description: Count of participants for whom there was an unintended dural puncture after placement
Time Frame: within 60min of first attempt at placement
Measure: Count of Participants; unit: Participants
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
Participants | 0 | 1
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p = 1.0000, Chi-squared

4. Secondary Outcome: Incidence of Paresthesia
Description: Count of participants for whom there was an incidence of paresthesia
Time Frame: within 60min of first attempt at placement
Measure: Count of Participants; unit: Participants
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
Participants | 8 | 4
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p = 0.3753, Chi-squared

5. Secondary Outcome: Incidence of Epidural Intravascular Cannulations
Description: Count of participants for whom there was an incidence of epidural intravascular cannulation
Time Frame: within 60min of first attempt at placement
Measure: Count of Participants; unit: Participants
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
Participants | 1 | 1
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p = 1.0000, Chi-squared

6. Secondary Outcome: Epidural Needle Manipulations Needed to Successfully Advance
Description: For each participant, the number of total manipulations (major or minor) needed to successfully advance catheter
Time Frame: within 60min of first attempt at placement
Measure: Count of Participants; unit: Participants
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
Number analyzed (Participants) | 120 | 120
Participants
  0 manipulations | 81 | 117
  1 manipulation | 19 | 2
  2 manipulations | 6 | 0
  3 manipulations | 6 | 0
  4 manipulations | 5 | 0
  5 manipulations | 2 | 1
  6 manipulations | 1 | 0
Statistical Analysis 1: Comparison: Arrow Catheter Kit. vs B.Braun Catheter Kit; Test type: Superiority; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Within 60 minutes of first attempt at placement
Arm/Group | Arrow Catheter Kit. | B.Braun Catheter Kit
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03722446/Prot_SAP_000.pdf